CLINICAL TRIAL: NCT04619810
Title: "Impact of a Nursing Intervention in the Management of Oncological Patients With Lung Cancer Under Treatment With Immunotherapy"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-IIE-2020-77
Record Dates: First submitted 2020-09-21; First posted 2020-11-06 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer
Keywords: immunotherapy; lung cancer; nurse intervention program
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other): quasi-experimental pre-post study
  Interventions: Other: Nurse intervention program

INTERVENTIONS:
Other: Nurse intervention program — Implementation of a specific care program for patients receiving immunotherapy for lung cancer

SUMMARY:
Introduction. Lung cancer is very common worldwide with 2.09 million cases in 2018. Immunotherapy has become a mainstay in cancer treatment. There is insuficient knowledge about the impact of altered needs, as well as the interventions developed by the nurse that are aimed at cancer patients in immunotherapy treatment.

Objectives. Describe the needs of non-microcytic lung cancer patients in immunotherapy. And, evaluate the effectiveness of a nurse intervention program aimed at these patients in decreasing comorbidities, increasing satisfaction, early detection of symptoms and management of toxicities, quality of life and monitoring of anthropometric indicators.

Methodology. Phase 1: descriptive, cross-cutting and prospective study. Phase 2: quasi-experimental pre-post study. The sample is patients of the Hospital de la Santa Creu i Sant Pau, with non-microcytic lung cancer in treatment with Checkpoints inhibitor antibodies. The dependent variables: sociodemographic variables, clinical variables, satisfaction, quality of life, nutritional status, psychological impact, toxicities, number of unscheduled visits and health costs. Independent variable: nurse intervention program.

Implications for practice: Knowing the needs of patients in immunotherapy treatment will allow the development of a nurse care program to meet these needs and evaluate the program.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (> or equal to 18 years), either male or female.
* Patient diagnosed with lung cancer regardless of subtype and / or stage. Except for small cell lung cancer, since this subtype of lung cancer is very different from the others and requires its own study.
* Patient receiving immunotherapy regardless of the treatment line.
* Patient who receives immunotherapy regardless of whether it is monotherapy or combination of chemotherapy.
* Patient who is able to consent to participate in the study.
* Patient who can read, understand and can communicate verbally.

Exclusion Criteria:

* Patient diagnosed with lung cancer synchronously with another neoplasm.
* Patients with speech disorders.
* Patients who do not understand or speak Spanish, Catalan or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Number of altered needs of patients with lung cancer undergoing treatment with immunotherapy | one day
  Detect the altered needs of patients with lung cancer in immunotherapy treatment. In order to outline the best intervention program that suits their needs. Through assessment through scales and questionnaires.
Changes on anxiety in lung cancer patients with immunotherapy treatment measured by Hospital Anxiety and Depression Scale (HADS) | 6 months
  Assess the patient's level of anxiety from diagnosis and prior to initiating treatment up to 6 months after initiating treatment. Using the Hospital Anxiety and Depression Scale (HADS)
Changes on quality of life in lung cancer patients with immunotherapy treatment measured by EORTC quality of life scale | 6 months
  Assess the quality of life of lung cancer patients from before starting immunotherapy up to 6 months after starting it. Through the EORTC QLQ-LC 30.
Number of immunomediated toxicities requiring hospital admission | 6 months
  Record the number and type of toxicities that require hospital admission for its management.

SECONDARY OUTCOMES:
Number of nutritional alterations in patients with lung cancer, who start immunotherapy treatment | 6 months
  Through the Nutriscore scale and to records of specific values of the blood analysis of the nutritional status of patients with lung cancer before starting immunotherapy and 6 months after starting it.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Jorgina Serra López, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Serra-Lopez J, Pujol-Besora C, Martinez-Recio S, Barba A, Riudavets Melia M, Sullivan I, Torralbas-Ortega J, Llado-Jordan G, Majem M, Martinez-Momblan MA. Clinical and economic impact of the advanced practice nurse in lung cancer patients receiving immunotherapy-based treatments: A quantitative study. Eur J Oncol Nurs. 2025 Feb;74:102809. doi: 10.1016/j.ejon.2025.102809. Epub 2025 Jan 23. PMID 39892201